CLINICAL TRIAL: NCT02788708
Title: Phase I Evaluation of Lenvatinib and Weekly Paclitaxel in Patients With Recurrent Endometrial, Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Lenvatinib and Weekly Paclitaxel for Patients With Recurrent Endometrial or Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Floor Backes (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor-Investigator, Floor Backes, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-15273; NCI-2016-00256 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-04-04; First posted 2016-06-02 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Fallopian Tube Carcinoma; Recurrent Ovarian Cancer; Primary Peritoneal Carcinoma; Recurrent Endometrial Cancer
Keywords: paclitaxel; lenvatinib
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms | interventions — lenvatinib; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenvatinib, paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and lenvatinib mesylate PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenvatinib Mesylate; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Drug: Lenvatinib Mesylate — Given PO
  Other Names: 4-[3-Chloro-4-(N'-cyclopropylureido)phenoxy]7-methoxyquinoline-6-carboxamide Mesylate; E7080; Multi-Kinase Inhibitor E7080
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of lenvatinib mesylate when given together with paclitaxel in treating patients with endometrial, ovarian, fallopian tube, or primary peritoneal cancer that has come back or grown. Lenvatinib mesylate may stop the growth of tumor cells by blocking a protein needed for cell growth and may block the growth of new blood vessels necessary for tumor growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving lenvatinib mesylate and paclitaxel together may work better in treating patients with endometrial, ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RPTD) of combination lenvatinib mesylate (lenvatinib) and weekly paclitaxel in patients with recurrent endometrial, epithelial ovarian, primary peritoneal, or fallopian tube carcinoma.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of combination lenvatinib and weekly paclitaxel in patients with recurrent endometrial, epithelial ovarian, primary peritoneal, or fallopian tube carcinoma.

II. To explore the objective antitumor activity (complete and partial response) of combination lenvatinib and weekly paclitaxel as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

III. To measure the progression free survival. IV. To evaluate the pharmacokinetics of combination paclitaxel and lenvatinib.

OUTLINE: This is a dose -escalation study of lenvatinib mesylate.

Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 and lenvatinib mesylate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed endometrial cancer, epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (all histological subtypes)who have disease progression after treatment with available therapies that are known to confer clinical benefit or who are intolerant to prior treatment
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral computerized tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have received prior treatment with a platinum containing regimen and may have received an unlimited number of prior regimens (including prior taxanes)
* Patients with ovarian, Fallopian tube or primary peritoneal cancer must be platinum resistant (progression < 6 months after completion of a platinum containing regimen)
* Patients may have received prior targeted therapy such as bevacizumab
* Eastern Cooperative Oncology Group performance status =< 1
* Leukocytes >= 3,000/mcL (microliter)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >=8.0 g/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Creatinine < 1.5 mg/dL X ULN OR creatinine clearance >= 30 mL/min for patients with creatinine levels above institutional normal
* Urine protein by dipstick <1+ or UPC =< 1.0 by urinalysis
* Patients with chronic hypertension that is well controlled with systolic blood pressure of < 140 mmHg or diastolic blood pressure of < 90 mmHg, and in whom there has been no change in blood pressure medication in the last two weeks, are eligible
* Patients who have a history of deep vein thrombosis (DVT) or pulmonary embolus and are stable on anticoagulation for > 1 month are eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of lenvatinib mesylate when given with paclitaxel defined as the highest dose level with =< 1 dose limiting toxicities among 6 patients graded by CTCAE | 4 weeks

SECONDARY OUTCOMES:
Objective antitumor activity (complete and partial response) assessed by RECIST criteria | Up to 5 years
Pharmacokinetics (PK) of combination paclitaxel and lenvatinib mesylate | Cycle 1 Day 1 and Day 15 (cycle is 28 days).
  Effect of lenvatinib on the pharmacokinetics of paclitaxel as well as the effect of paclitaxel on the pharmacokinetics of lenvatinib will be studied. Plasma samples will be collected on Cycle 1, Day 1 and Day 15.
Progression free survival | months

CONTACTS AND LOCATIONS:
Overall Officials: Floor Backes, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu